CLINICAL TRIAL: NCT05023421
Title: Investigation of the Relationship Between the Use of Social Media and Gross Motor Function, Hand Function, Communication, Eating and Drinking and Visual Function Children With Cerebral Palsy in Turkey.
Brief Title: Investigation of the Relationship Between the Use of Social Media and Functional Level in Children With CP
Acronym: IRoSMFLCP
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Mintaze Kerem Gunel, Professor, Phd, Hacettepe University
Other Study IDs: GO: 20/450
Record Dates: First submitted 2021-08-07; First posted 2021-08-26 (Actual); Last update posted 2021-08-26 (Actual); Status verified 2021-08

CONDITIONS: Social Media Addiction; Cerebral Palsy
Keywords: problematic media use; cerebral palsy; physical therapy; motor function
MeSH Terms: conditions — Internet Addiction Disorder; Cerebral Palsy

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Problematic media use of children with CP: The participants in the current study were parents of children with CP aged 4-18 years. They were recruited at the Hacettepe University Physical Therapy and Rehabilitation Faculty Cerebral Palsy and Pediatric Rehabilitation Unit and Special Education and Rehabilitation Centers. The inclusion criteria were having a child with CP aged 2-18 years without severe cognitive problems, being a primary caregiver.
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
The aim of this study is to examine the relationship between screen usage time and problematic social media use in children with Cerebral Palsy (CP) with motor function, hand function, speech and vision function.

DETAILED DESCRIPTION:
Problematic Media Use Measure, Strengths and Difficulties Questionnaire were administered to 158 parents of children with CP. In order to determine the screen usage time, parents were asked about the screen usage time of their children on weekdays and weekends, and the average usage time in a week was calculated. Gross Motor Function Classification System (GMFCS), Manual Abilities Classification System (MACS), Eating and Drinking Ability Classification System (EDACS), Communication Function Classification System (CFCS),and Visual Function Classification System (VFCS) were used to determine functional levels.The structural equation model was used for statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Parents of children with CP aged 4-18 years
* Parents of children with CP without severe cognitive problems, being a primary caregiver.

Exclusion Criteria:

* Not being a primary caregiver

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The participants in the current study were parents of children with CP aged 4-18 years.
  The inclusion criteria were having a child with CP aged 2-18 years without severe cognitive problems, being a primary caregiver.
Sampling Method: Probability Sample
Enrollment: 158 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Problematic Media Use Measure | At baseline
  Problematic Media Use Measure (PMUM) was developed by Domoff et al. to detect problematic media use in children aged 4-11. Both the long form and the short form of the scale have only one factor structure. Items are scored on a Likert scale from 1 (never) to 5 (always). PMUM total score is obtained by taking the average of scores from all items. High scores from the scale indicate problematic use. The scale, which is applied by parents considering behavior of the child, tries to detect not the problematic use of a specific media tool, but generally the problematic use of visual media tools (such as television, computer, tablet, phone), in other words, screen addiction.

SECONDARY OUTCOMES:
Strength and Difficulties Questionniare | At baseline
  Strength and Difficulties Questionniare (SDQ) is used to screen emotional and behavioral problems. The scale, which consists of 25 items in total, has 5 sub-dimensions: attention deficit and hyperactivity, behavioral problems, emotional problems, peer problems and social behaviors. Scale scoring was made as "0 (not correct)", "1 (partially correct)", "2 (absolutely correct)" for each statement. Turkish validity and reliability study has been done

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Eyalet/Yerleşke, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No